CLINICAL TRIAL: NCT06342544
Title: Immediate Corticosteroid Therapy and Rituximab to Prevent Generalization in Ocular Myasthenia: a PROBE Multicenter Open-label Randomized Controlled Trial.
Acronym: IMCOMG
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AGN_2023_14
Record Dates: First submitted 2024-03-22; First posted 2024-04-02 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Ocular Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate treatment with corticosteroids addition of rituximab if recurrence (Experimental)
  Interventions: Drug: immediate treatment with corticosteroids; Drug: addition of rituximab if recurrence
- based on standard practice (No Intervention)

INTERVENTIONS:
Drug: immediate treatment with corticosteroids — Immediate standardized treatment with corticosteroids. Standardized treatment in the experimental arm will start at 0.5mg/kg/d prednisone.
  Arms: immediate treatment with corticosteroids addition of rituximab if recurrence
Drug: addition of rituximab if recurrence — rituximab added if ocular symptoms reappear as corticosteroids are tapered off. Rituximab will be given at a dose of 500mg/6months for 12 months.
  Arms: immediate treatment with corticosteroids addition of rituximab if recurrence

SUMMARY:
Myasthenia is an autoimmune disease causing dysfunction of the neuromuscular junction, resulting in fluctuating and variable muscle weakness.

In the initial phase of the disease, 70% of patients present with ocular onset myasthenia (OMG), i.e. weakness limited to the oculomotor muscles. Generalization to skeletal, bulbar and axial muscles occurs in 20-40% of cases, with a higher frequency in the first and second years, respectively 46% and 60% of generalizations. This reflects the maturation of the autoimmune response in the early years of the disease, and represents a therapeutic window of opportunity to modify the course of the disease.

Generalization is a critical event, putting the patient at risk of admission to an intensive care unit and necessitating the use of long-term immunosuppressants.

There is currently no validated strategy for preventing generalization. On the one hand, a preventive role for corticosteroid therapy in ocular-onset myasthenia has been observed in some studies, but not confirmed by others. These contradictory results may be explained by the bias of retrospective observational studies and the use of different corticosteroid administration regimens.

On the other hand, recent data on the use of low-dose Rituximab in the early phase of the disease shows greater efficacy than later use, enabling prolonged remission of the disease with a very good tolerability profile.

We propose to compare in a randomized controlled trial the usual practice with a proactive strategy with a standardized corticosteroid regimen immediate at diagnosis.

Patients with ocular myasthenia are usually treated symptomatically with acetylcholinesterase inhibitors. The introduction of corticosteroids is delayed and limited to patients with persistent disabling diplopia or ptosis with occlusion. When corticosteroids are tapered off, ocular symptoms may recur. This level of corticosteroid dependence observed in patients treated for ocular myasthenia has not been specifically studied. In order to reduce the levels of corticosteroids administered and avoid recurrence of ocular symptoms and their delayed generalization, it is usually proposed to introduce another immunosuppressant.

The aim of this study is to evaluate the efficacy of a standardized proactive prevention strategy on the generalization of ocular onset myasthenias during the first 2 years. It will combine immediate treatment with corticosteroids at the time of diagnosis, with the addition of rituximab in the event of recurrence of ocular symptoms as corticosteroids are tapered off.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Diagnosis of ocular myasthenia within the last 6 months, defined :

  * either by a typical clinical examination objectified by an expert clinician: ptosis and/or binocular diplopia, with a variable and fluctuating character (either spontaneous or provoked by effort or rest)
  * or by positive anti-AChR antibodies or the presence of decrement on repetitive nerve stimulation or a positive edrophonium test
* Ocular symptoms lasting at least one month and limited to extra-ocular muscles (weakness in one or both orbicularis oculi)
* No non-ocular symptoms on MMS, MGC and MG-ADL.
* Naïve to immunosuppressive therapy for ocular myasthenia gravis.

Exclusion Criteria:

* Thymoma
* Pupillary anomaly other than that resulting from previous local disease or surgery.
* Signs of restrictive abduction or supraduction myopathy due to dysthyroid ophthalmopathy.
* Graves' ophthalmopathy
* Onset of ocular symptoms more than one year before screening date
* Hypersensitivity to rituximab, murine proteins, prednisone, methylprednisone, aziathioprine or 6-mercaptopurine, paracetamol, dexchlorpheniramine.
* Any infectious condition
* Patients with severe immune deficiency
* Severe heart failure (New York Heart Association (NYHA) Class IV) or severe uncontrolled heart disease
* Severe hepatic insufficiency
* Psychotic states not yet controlled by treatment
* Hyperuricemia on xanthine oxidase inhibitors (allopurinol and febuxostat)
* Risk of angle-closure glaucoma
* Risk of urinary retention due to urethro-prostatic disorders
* Vaccination with live attenuated vaccine required during study and up to 6 months after rituximab discontinuation
* Women of childbearing age who do not wish to use effective contraception during their participation and at least 12 months after
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
proportion of patients who progressed to generalized myasthenia within 2 years of follow-up | Day0 to month24
  Generalization is defined by a loss of 5 points or more on any Myasthenic Muscle Score (MMS) item, excluding "eyelid occlusion" and "extrinsic ocular musculature".
  Progress towards generalization will be assessed by an expert physician, blinded to the intervention arm.

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - Centre Hospitalier Universitaire De Bordeaux, Bordeaux
  - Hôpital Raymond Pointcarre, Garches
  - Centre Hospitalier Universitaire De Lille, Lille
  - Hospices Civils De Lyon, Lyon
  - Centre Hospitalier Universitaire De Nice, Nice
  - CHNO, Paris
  - Hôpital de la Pitié-Salpêtrière, Paris
  - Centre Hospitalier Sainte Anne, Paris
  - Fondation Adolphe de Rothschild, Paris
  - Les Hopitaux Universitaires De Strasbourg, Strasbourg
  - Centre Hospitalier Universitaire De Toulouse, Toulouse